CLINICAL TRIAL: NCT03939533
Title: Clinical Phase 3 Study to Monitor the Safety, Tolerability, and Efficacy of Subcutaneous Human Immunoglobulin (CUTAQUIG®) Administered at Modified Dosing Regimens in Patients With Primary Immunodeficiency Diseases
Brief Title: Study to Monitor Subcutaneous Human Immunoglobulin Administered at Modified Dosing Regimens in Patients With Primary Immunodeficiency Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCGAM-06
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Primary Immune Deficiency Disorder
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Increased Volume Cohort - Cohort 1 (Experimental): Increased volume at each infusion site - patients will receive CUTAQUIG weekly and increase infusion volumes every 4 weeks
  Interventions: Drug: CUTAQUIG
- Increased Infusion Rate Cohort - Cohort 2 (Experimental): Increased infusion rate - patients will receive CUTAQUIG weekly and increase infusion rates every 4 weeks
  Interventions: Drug: CUTAQUIG
- Every Other Week Dosing Cohort - Cohort 3 (Experimental): Every other week dosing - patients will receive CUTAQUIG every other week at the equivalent of twice their body-weight dependent [mg/kg] weekly dose
  Interventions: Drug: CUTAQUIG

INTERVENTIONS:
Drug: CUTAQUIG — Human normal immunoglobulin

SUMMARY:
CLINICAL PHASE 3 STUDY TO MONITOR THE SAFETY, TOLERABILITY, AND EFFICACY OF SUBCUTANEOUS HUMAN IMMUNOGLOBULIN (CUTAQUIG®) ADMINISTERED AT MODIFIED DOSING REGIMENS IN PATIENTS WITH PRIMARY IMMUNODEFICIENCY DISEASES

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥2 years and ≤75 years.
2. Confirmed diagnosis of primary immunodeficiency (PI) disease as defined by the European Society for Immunodeficiencies and Pan American Group for Immunodeficiency and requiring immunoglobulin replacement therapy due to hypogammaglobulinaemia or agammaglobulinaemia. Note: The exact type of PI disease will be recorded.
3. Established on a consistent or stable mg/kg dose of any SCIG treatment for a minimum of 3 months prior to Screening. Note: patients entering Cohort 3 must be on weekly SCIG infusions for a minimum of 12 weeks.
4. Availability of the Immunoglobulin G (IgG) trough levels of 2 previous SCIG infusions within 1 year of Screening, with 1 trough level obtained within 3 months prior to enrollment, and maintenance of trough serum IgG levels

   ≥5.0 g/L in 2 previous infusions. Patients with no prior IgG trough level within 3 months prior to enrollment may use the Screening IgG trough level as their 2nd reading.
5. Voluntarily given, fully informed signed informed consent. For patients under the legal age of consent, voluntarily given, fully-informed, signed informed consent will be provided by patient's parent or legal guardian, and assent will be provided by patient (per age-appropriate Institutional Review Board [IRB] requirements).
6. Females of childbearing potential, who are not nursing and have no plans for pregnancy during the course of the study, have been using at least 1 acceptable form of birth control for a minimum of 30 days prior to the Screening visit and must agree to use at least 1 acceptable method of contraception for 30 days after the last dose of CUTAQUIG. Acceptable methods include: intrauterine device (IUD), hormonal contraception, male or female condom, spermicide gel, diaphragm, sponge, cervical cap, or abstinence.
7. For female patients of child-bearing potential, a negative result in a urine pregnancy test conducted at the Screening visit.
8. Willingness to comply with all aspects of the protocol, including blood sampling, for the duration of the study.

Exclusion Criteria:

1. Evidence of active infection within 4 weeks of Screening or during the Screening Period.
2. Current or clinically-significant history of any cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological (excluding PI), hematologic, and/or psychiatric disorder(s), or a history of any other illness that, in the opinion of the Investigator, might confound the results of the study, or pose additional risk to the patient by participation in the study.
3. Known history of adverse reactions to immunoglobulin A (IgA) in other products.
4. Body mass index (BMI) >40 kg/m2 for patients entering Cohort 2 or Cohort 3. There are no BMI restrictions for Cohort 1.
5. Ongoing history of hypersensitivity or persistent reactions to blood or plasma derived products, or any component of the investigational product (such as Polysorbate 80).
6. Requirement of any routine premedication for IgG administration.
7. History of malignancies of lymphoid cells and immunodeficiency with lymphoma.
8. Severe liver function impairment (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >3 times above upper limit of normal).
9. Known protein-losing enteropathies or clinically significant proteinuria.
10. Presence of renal function impairment (creatine >120 μM/L or creatinine >1.35 mg/dL), or predisposition for acute renal failure (eg, any degree of preexisting renal insufficiency or routine treatment with known nephritic drugs).
11. Treatment with oral or parenteral steroids for ≥30 days, or when given intermittently or as bolus at daily doses ≥0.15 mg/kg when taken within 30 days of Screening. Note: Short or intermittent courses of steroids (ie, a steroid burst) of >0.15 mg/kg/day is allowed for treatment of a short-term condition such as an asthma exacerbation.
12. Treatment with immunosuppressive or immunomodulatory drugs (except Omalizumab).
13. Use of HYQVIA (Immune Globulin Infusion 10% [Human] with Recombinant Human Hyaluronidase) within 3 months prior to first CUTAQUIG infusion.
14. Live viral vaccination (such as measles, rubella, mumps, and varicella) within 2 months prior to first CUTAQUIG infusion.
15. Exposure to blood or any blood product or derivative, other than subcutaneous IgG used for regular PI disease treatment, within 3 months before the first CUTAQUIG infusion.
16. Treatment with any investigational medicinal product within 3 months prior to first CUTAQUIG infusion. Note: Patients participating in Study SCGAM-03 will be allowed to enter this study without the 3-month waiting period for an Investigational Product. Patients receiving another SCIG product within 3 months prior to the first CUTAQUIG infusion may be considered for enrollment after Sponsor approval.
17. Presence of any condition that is likely to interfere with the evaluation of CUTAQUIG or satisfactory conduct of the trial.
18. Known or suspected to abuse alcohol, drugs, psychotropic agents, or other chemicals within the past 12 months prior to first CUTAQUIG infusion.
19. Known active or chronic hepatitis B, hepatitis C, or HIV infection. Past hepatitis B or hepatitis C infection that has been cured is allowed.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Octapharma Research Site, Scottsdale, Arizona
  - Octapharma Research Site, Irvine, California
  - Octapharma Research Site, Santa Barbara, California
  - Octapharma Research Site, Centennial, Colorado
  - Octapharma Research Site, North Palm Beach, Florida
  - Octapharma Research Site, St. Petersburg, Florida
  - Octapharma Research Site, Albany, Georgia
  - Octapharma Research Site, Louisville, Kentucky
  - Octapharma Research Site, Chevy Chase, Maryland
  - Octapharma Research Site, St Louis, Missouri
  - Octapharma Research Site, Papillion, Nebraska
  - Octapharma Research Site, Asheville, North Carolina
  - Octapharma Research Site, Cincinnati, Ohio
  - Octapharma Research Site, Mayfield, Ohio
  - Octapharma Research Site, Toledo, Ohio
  - Octapharma Research Site, Pittsburgh, Pennsylvania
  - Octapharma Research Site, Dallas, Texas
  - Octapharma Research Site, Bellingham, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with a history of primary immunodeficiency (PI) disease that were currently on a stable does of SCIG treatment were enrolled at 16 research sites across the US between October 2019 and January 2022
Period: Overall Study
Arm/Group | Increased Volume Cohort - Cohort 1 | Increased Infusion Rate Cohort - Cohort 2 | Every Other Week Dosing Cohort - Cohort 3
Started | 15 | 15 | 34
Completed | 12 | 13 | 30
Not Completed | 3 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Increased Volume Cohort - Cohort 1 | Increased Infusion Rate Cohort - Cohort 2 | Every Other Week Dosing Cohort - Cohort 3 | Total
Number analyzed (Participants) | 15 | 15 | 34 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.20 (17.27) | 47.88 (20.53) | 50.81 (18.54) | 50.21 (18.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 27 | 48
  Male | 5 | 4 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 12 | 15 | 34 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0
Type of PI Disease [Count of Participants; unit: Participants] — Primary Immunodeficiency Disease type of enrolled subjects
  Participants
    Common Variable Immunodeficiency (CVID) | 14 | 13 | 30 | 57
    X-linked Agammaglobulinemia (XLA) | 0 | 1 | 0 | 1
    Other | 1 | 1 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: IgG Trough Levels From Baseline to End of Study (28 Weeks)
Description: Mean change from baseline in individual total IgG trough levels in cohort 3 from weekly infusions to end of study (28 weeks) every other week infusions, and for cohort 1 and cohort 2 (weekly infusions) change from baseline through study completion (28 weeks)
Time Frame: Through study completion, up to 28 weeks
Population: Cohort 3
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Increased Volume Cohort - Cohort 1; Increased Infusion Rate Cohort - Cohort 2: Increased infusion rate - patients will receive CUTAQUIG weekly and increase infusion rates every 4 weeks
  CUTAQUIG: Human normal immunoglobulin
Arm/Group | Increased Volume Cohort - Cohort 1 | Increased Infusion Rate Cohort - Cohort 2 | Every Other Week Dosing Cohort - Cohort 3
Number analyzed (Participants) | 15 | 15 | 31
g/L | 0.144 (0.7303) | 0.065 (1.1046) | -0.593 (1.0791)

2. Secondary Outcome: Serious Bacterial Infection Rates
Description: Number of subjects who reported SBIs during the study
Time Frame: Through study completion, up to 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Increased Volume Cohort - Cohort 1 | Increased Infusion Rate Cohort - Cohort 2 | Every Other Week Dosing Cohort - Cohort 3
Number analyzed (Participants) | 15 | 15 | 34
Participants | 0 | 0 | 0

3. Secondary Outcome: Time to Resolution of Infections
Description: The amount of days it took for infectious disease occurrence and resolution for subjects
Time Frame: Through study completion, 28 weeks
Measure: Median (Full Range); unit: days
Arm/Group | Increased Volume Cohort - Cohort 1 | Increased Infusion Rate Cohort - Cohort 2 | Every Other Week Dosing Cohort - Cohort 3
Number analyzed (Participants) | 15 | 15 | 34
days | 23.5 [1 to 160] | 20.0 [11 to 85] | 16.0 [6 to 65]

4. Secondary Outcome: Antibiotic Usage
Description: Amount of subjects treated with antibiotics during the study
Time Frame: Through study completion, up to 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Increased Volume Cohort - Cohort 1 | Increased Infusion Rate Cohort - Cohort 2 | Every Other Week Dosing Cohort - Cohort 3
Number analyzed (Participants) | 15 | 15 | 34
Participants | 10 | 8 | 21

5. Secondary Outcome: Number of Antibiotic Treatment Episodes Annualized
Description: Total number of treatment episodes annualized calculated as the sum of all unique episodes of antibiotics of all subjects from first dose day of cutaquig to last study visit/number of person years exposure
Time Frame: Through study completion, up to 28 weeks
Measure: Number; unit: episodes per person year
Arm/Group | Increased Volume Cohort - Cohort 1 | Increased Infusion Rate Cohort - Cohort 2 | Every Other Week Dosing Cohort - Cohort 3
Number analyzed (Participants) | 15 | 15 | 34
episodes per person year | 4.53 | 1.96 | 2.38

ADVERSE EVENTS:
Time Frame: Through study complete, up to 28 weeks
Arm/Group | Increased Volume Cohort - Cohort 1 | Increased Infusion Rate Cohort - Cohort 2 | Every Other Week Dosing Cohort - Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 1/34
Other Adverse Events (participants affected / at risk) | 13/15 | 12/15 | 30/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Increased Volume Cohort - Cohort 1 (N=15) | Increased Infusion Rate Cohort - Cohort 2 (N=15) | Every Other Week Dosing Cohort - Cohort 3 (N=34)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Increased Volume Cohort - Cohort 1 (N=15) | Increased Infusion Rate Cohort - Cohort 2 (N=15) | Every Other Week Dosing Cohort - Cohort 3 (N=34)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (9) | 2 (5)
Fatigue (General disorders) | 2 (2) | 1 (7) | 1 (1)
Infusion Site Erythema (General disorders) | 4 (7) | 8 (54) | 8 (12)
Infusion Site Pain (General disorders) | 2 (2) | 4 (10) | 3 (7)
Infusion Site Pruritis (General disorders) | 4 (15) | 5 (19) | 6 (10)
Pyrexia (General disorders) | 1 (1) | 1 (4) | 2 (3)
Acute Sinitus (Infections and infestations) | 2 (2) | 2 (3) | 2 (2)
Ear Infection (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 4 (4) | 5 (8) | 6 (9)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Heachache (Nervous system disorders) | 0 (0) | 3 (4) | 7 (16)

LIMITATIONS AND CAVEATS:
For outcome #3, 'Mean' is correct. The values presented are indeed calculated as means using the usual formula (only for the CIs a compound Poisson process model is used to account for the intra-patient correlation in incidents).For each patient, the annual infection rate was calculated as # of infections/observation period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT03939533/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT03939533/SAP_001.pdf